CLINICAL TRIAL: NCT07081022
Title: JS203 Combination Regimens in B-Cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS203-002-II-B-NHL
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Gemcitabine; Oxaliplatin; Ifosfamide; Carboplatin; Etoposide; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- DLBCL-Gemox (Experimental): In participants with relapsed/refractory diffuse large B cell lymphoma ineligible for ASCT
  Interventions: Drug: JS203 in combination with gemcitabine and oxaliplatin
- DLBCL-ICE (Experimental): In participants with relapsed/refractory diffuse large B cell lymphoma intended for ASCT
  Interventions: Drug: JS203 in combination with ifosfamide, carboplatin and etoposide
- DLBCL- RCHOP (Experimental): In participants with newly diagnosed diffuse large B cell lymphoma
  Interventions: Drug: JS203 in combination with rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone
- FL-Lena (Experimental): In participants with relapsed/refractory follicular lymphoma
  Interventions: Drug: JS203 combined with lenalidomide
- MCL-Lena (Experimental): In participants with relapsed/refractory mantle cell lymphoma
  Interventions: Drug: JS203 combined with lenalidomide
- MZL-Lena (Experimental): In participants with relapsed/refractory marginal zone lymphoma
  Interventions: Drug: JS203 combined with lenalidomide

INTERVENTIONS:
Drug: JS203 in combination with gemcitabine and oxaliplatin — Gemcitabine and oxaliplatin 8 cycles (Q3W) and JS203 (21 days/cycle) Cycle 1 QW,Cycle 2 and therafter Q3W until progression or unacceptable toxicity.
  Arms: DLBCL-Gemox
Drug: JS203 in combination with ifosfamide, carboplatin and etoposide — Ifosfamide, carboplatin and etoposide, 3 cycles (Q3W) and JS203, Cycle 1 QW, Cycle 2 and therafter Q3W until trasnplant, progression or unacceptable toxicity.
  Arms: DLBCL-ICE
Drug: JS203 in combination with rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone — Rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone 6 cycles (Q3W) and JS203, 8 cycles (21 days/cycle), Cycle 1 QW, Cycle 2 to Cycle 8 Q3W.
  Arms: DLBCL- RCHOP
Drug: JS203 combined with lenalidomide — lenalidomide,12 cycles, Cycle 1(Q3W), Cycle 2 to Cycle 12 (Q4W) and JS203, 12 cycles, Cycle 1 (21 days/cycle) QW, Cycle 2 to Cycle 12 (28 days/cycle) Q4W.
  Arms: FL-Lena; MCL-Lena; MZL-Lena

SUMMARY:
To evaluate the preliminary efficacy of JS203 combined with standard regimens in patients with B-cell Non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled：

* Age range: 18 to 80 years old (inclusive), both male and female are acceptable；
* ECOG: 0-2；
* B-cell non-Hodgkin's lymphoma expressing CD20 antigen that has been pathologically diagnosed；
* At least one measurable lesion meeting the criteria specified in the Lugano 2014 response assessment； Acceptable organ function at screening；

Exclusion Criteria:

* A history of severe allergy to monoclonal antibody therapy (or recombinant antibody-related fusion protein)；
* Previously received CD20-CD3 bispecific antibody treatment；
* Previous allogeneic hematopoietic stem cell transplantation；
* Previous solid organ transplantation；
* History of autoimmune diseases；
* Patients with a history of macrophage activation syndrome (MAS)/ hemophagocytic lymphohistiocytosis (HLH)；
* Patients with a history of progressive multifocal leukoencephalopathy (PML)；
* A known or suspected history of CNS lymphoma (including primary or secondary)；
* There is pleural effusion, peritoneal effusion or pericardial effusion that requires treatment (such as puncture or drainage)；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 15 months
  Objective response rate (ORR) based on 2014 Lugano criteria

SECONDARY OUTCOMES:
complete response (CR) | up to approximately 24 months
  The complete response rate (CR) evaluated based on 2014 Lugano criteria
Duration of response (DoR) | up to approximately 24 months
  Duration of response (DoR) evaluated based on 2014 Lugano criteria
Duration of complete response (DoCR) | up to approximately 24 months
  Duration of complete response (DoCR) evaluated based on 2014 Lugano criteria
Time to response (TTR) | up to approximately 24 months
  Time to response (TTR) evaluated based on 2014 Lugano criteria
Progression-free survival (PFS) | up to approximately 24 months
  Progression-free survival (PFS) evaluated based on 2014 Lugano criteria
Overall survival (OS) | up to approximately 24 months
  Overall survival (OS) evaluated based on 2014 Lugano criteria
Adverse events (AE) | up to approximately 24 months
  Incidence and severity of all adverse events (AE) that occurred during the clinical trial
PK | up to approximately 24 months
  The serum drug concentration of JS203
ADA | up to approximately 24 months
  The incidence and titer of the anti-drug antibody (ADA) of JS203
NAb | Up to approximately 24 months
  The incidence of neutralizing antibodies (NAb) of JS203 (if applicable)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No